CLINICAL TRIAL: NCT05447325
Title: Neuroimaging Approaches to Improve Prediction of Smoking Initiation and Nicotine Use Escalation Among Young Adult Electronic Nicotine Delivery Systems Users
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Jiaying Liu, Associate Professor, University of Georgia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PROJECT00003494
Record Dates: First submitted 2022-05-01; First posted 2022-07-07 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Message Exposure (Sequence: Regular Then Flavor); Message Exposure (Sequence: Flavor Then Regular); No Message Exposure (Control Condition)
Keywords: health message intervention; randomized controlled trial

STUDY DESIGN:
Intervention Model Description: In the PSA exposure conditions, half of the participants will receive regular PSA exposure during the first 6 months and then switch to receiving flavor PSA exposure during the second 6 months; the other half will first receive flavor PSAs, and then the regular PSAs.
Who Masked: Participant
Masking Description: The participants will be prevented from having knowledge of the interventions assigned to them.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Message exposure (sequence: regular PSAs then flavor PSAs) (Experimental): Participants randomly assigned to this arm will receive weekly emails and text messages of regular PSAs (i.e., focused in general on the negative consequences of vaping) for the first 6 months of the study, and will then receive weekly emails and text messages of flavor PSAs (i.e., focused specifically on harms and negative consequences associated with vaping flavored e-cigarette products) for the second 6 months of the study.
  Interventions: Behavioral: Exposure to Anti-Vaping Messages (generic themes then flavor-specific themes)
- Message exposure (sequence: flavor PSAs then regular PSAs) (Experimental): Participants randomly assigned to this arm will receive weekly emails and text messages of flavor PSAs (i.e., focused specifically on harms and negative consequences associated with vaping flavored e-cigarette products) for the first 6 months of the study, and will then receive weekly emails and text messages of regular PSAs (i.e., focused in general on the negative consequences of vaping) for the second 6 months of the study.
  Interventions: Behavioral: Exposure to Anti-Vaping Messages (flavor-specific themes then generic themes)
- No message exposure (control condition) (Experimental): Participants will not be receiving any PSA exposure over the 12 months.
  Interventions: Behavioral: Exposure to Anti-Vaping Messages (no message exposure)

INTERVENTIONS:
Behavioral: Exposure to Anti-Vaping Messages (generic themes then flavor-specific themes) — Messages are in the format of public service announcement (PSA) images that contain both textual (1-2 brief sentences) and illustrative visual components. The messages are designed to educate the participants about the harms and costs associated with e-cigarette use (e.g., negative health consequences, undesirable social perceptions, etc.). Half of the messages focus specifically on the harms and costs associated with using flavored vape products, while the other half address vaping harms broadly (i.e., not specifically focus on those related to flavored vaping). Participants in this arm will receive anti-vaping messages through emails and text messages every week. Specifically, over the course of a year, during the first six months, they will receive generic/regular PSAs that address vaping harms more broadly; during the second six months, they will receive flavor-specific PSAs that address vaping harms specifically associated with the use of flavored vape products.
  Arms: Message exposure (sequence: regular PSAs then flavor PSAs)
Behavioral: Exposure to Anti-Vaping Messages (flavor-specific themes then generic themes) — Messages are in the format of public service announcement (PSA) images that contain both textual (1-2 brief sentences) and illustrative visual components. The messages are designed to educate the participants about the harms and costs associated with e-cigarette use (e.g., negative health consequences, undesirable social perceptions, etc.). Half of the messages focus specifically on the harms and costs associated with using flavored vape products, while the other half address vaping harms broadly (i.e., not specifically focus on those related to flavored vaping). Participants in this arm will receive anti-vaping messages through emails and text messages every week. Specifically, over the course of a year, during the first six months, they will receive flavor-specific PSAs that address vaping harms specifically associated with the use of flavored vape products; during the second six months, they will receive generic/regular PSAs that address vaping harms more broadly.
  Arms: Message exposure (sequence: flavor PSAs then regular PSAs)
Behavioral: Exposure to Anti-Vaping Messages (no message exposure) — Participants will not receive any message intervention in this arm.
  Arms: No message exposure (control condition)

SUMMARY:
180 young adult vapers who are not current smokers will participate in a baseline functional magnetic resonance imaging (fMRI) experiment, prospectively linked to a 1-year randomized controlled trial. Baseline fMRI tasks will probe critical neurocognitive markers with high potential to account for individual differences in nicotine use prognosis and responsiveness to anti-vaping public service announcements (PSAs). Participants will be assigned randomly to a survey-only control condition, or one of two intervention orders, Regular PSA then Flavor PSA, and Flavor PSA then Regular PSA (n=60 each) in a 1-year counterbalanced crossover design. Every week intervention groups will receive anti-vaping PSAs either do not specifically address harms associated with vaping flavors (regular PSAs) or PSAs with a theme focusing on the harms of flavored vape products (flavor PSAs). Participants of the intervention groups will switch PSA exposure condition after 6 months. Their evaluations of the PSAs will be assessed with brief weekly online surveys. The links to the weekly online surveys will be sent via e-mail and text which allow them to access the surveys using any device with an internet browser. During the survey, the PSA of that week will first be displayed to PSA groups (n=120), followed by a query to provide message evaluation. Afterward, the survey questions will also assess their e-cigarette, cigarette, other tobacco use, and nicotine dependence, during the past week. The control group (n=60) will complete the surveys without viewing PSAs. In-person assessments at 3, 6, 9, and 12 months will biochemically confirm nicotine exposure.

DETAILED DESCRIPTION:
180 young adult current vapers will be recruited from multiple sources including the University of Georgia (UGA) student research pools from the Communication, Psychology, and Sociology Departments, posters, yard signs, local community liaisons, and via Craigslist and social media ads. The screening will begin with a brief online survey. The link to the survey will be included in the research pool websites, flyers, and social media ads. Those eligible after the screening will be invited to interview via Zoom for a more detailed assessment of eligibility. Eligible participants will be sent a pre-scan survey (about 0.5 hours) 24 hours prior to the in-person lab visit. They will then be invited to a 1.5-hour visit to UGA's Bioimaging Research Center (BIRC) and instructed to vape, or not, as usual that day. Upon arrival, participants' eligibility will be confirmed, and written informed consent will be obtained. Breath and urine samples will be collected to biochemically confirm the level of nicotine exposure (i.e., tobacco use severity), followed by the remaining pre-scan measures. Participants will then be trained to perform the fMRI tasks. During fMRI, they will wear earplugs and MR-compatible vision correction, if needed, and lie on the scanner table. Stimuli will be back-projected, and responses collected using a four-button response box configured to allow on-screen Likert scale ratings of 1-7, both via Eprime 3.0 software. MRI will last approximately 60min, followed by post-scan measures (about 0.5 hours).

After the baseline fMRI scan, investigators will deliver static, visual, and textual anti-vaping public service announcements (PSAs) and assess participants' evaluations of the PSAs weekly through brief online surveys via e-mails and text messages. In the two PSA conditions, every week participants will receive an email and a text message through which a static visual anti-vaping PSA will be displayed to them before a query to evaluate the perceived effectiveness of the PSAs, followed by questions about their tobacco use status during the past week. Half of the PSA condition participants (n=60) will be exposed to regular PSAs that focus generally on the negative consequences of vaping, and the other half (n=60) will be exposed to flavor PSAs, which focus specifically on the harms and negative consequences associated with vaping flavored e-cigarettes. Flavor PSAs will be both drawn from existing regular PSAs and created by adding a flavor theme on regular PSAs because existing flavor PSAs are still rare. PSA condition participants will switch types of PSA exposure after 6 months. Each week a different PSA will be displayed to the participants. Therefore, half of the PSA condition participants will be exposed to 24 regular PSAs during the first 6 months, and then to 24 flavor PSAs during the second 6 months. For the other half of the PSA condition participants, they will also be displayed the same 48 PSAs, but in the reverse sequence, i.e., 24 flavor PSAs first, then 24 regular PSAs next. Participants in the control condition (n=60) will directly answer the survey questions about their tobacco use status during the past week without PSA exposure and evaluation.

At 3-, 6-, 9- and 12-months participants will complete a 15-min visit that includes a CO confirmation for smoking, a urinary cotinine test for nicotine use, and other in-person follow-up measures.

ELIGIBILITY:
Inclusion Criteria:

* used e-cigarettes or other vaping devices at least 3 days during the past 30 days
* did not smoke a cigarette, even one or two puffs, during the past 30 days
* Magnetic resonance imaging (MRI) compatible and safe

Exclusion Criteria:

* used e-cigarettes or other vaping devices for less than 3 days during the past 30 days
* any use of cigarettes during the past 30 days
* history of a major neurological, psychiatric, or medical disorder
* MRI contraindications

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Self-report monthly smoking severity | 12 months
  The monthly number of cigarettes smoked will be assessed with the timeline follow-back measures. Specifically, participants will be asked to retrospectively estimate their daily cigarette use for the 7 days prior to the weekly survey date. The four weekly estimates will be averaged to create the monthly smoking severity measure. The greater the number, the higher the smoking severity in that month.
Self-report monthly vaping severity | 12 months
  The monthly number of vaping sessions (a vaping session refers to a minimum of about 15 puffs or vaping that lasts around 10 minutes) will be assessed with the timeline follow-back measures. Specifically, participants will be asked to retrospectively estimate their daily vaping sessions for the 7 days prior to the weekly survey date. The four weekly estimates will be averaged to create the monthly vaping severity measure. The greater the number, the higher the vaping severity in that month.
Exhaled carbon monoxide (CO) levels | 12 months
  Quarterly assessed exhaled CO levels quantified by parts per million (PPM)
Urine cotinine levels | 12 months
  Quarterly assessed urine cotinine levels (none, low, medium, high)

SECONDARY OUTCOMES:
Self-report monthly other tobacco use severity | 12 months
  Frequency of other tobacco use will be assessed by the timeline follow-back measures. Specifically, participants will be asked to retrospectively estimate their daily use of other tobacco for the 7 days prior to the weekly survey date. The four weekly estimates will be averaged to create the monthly other tobacco use severity measure. The greater the number, the higher the other tobacco use severity in that month.
Cigarette smoking urge | 12 months
  Levels of cigarette smoking will be assessed with the Brief Questionnaire of Smoking Urges (10 items;1= strongly disagree, 7= strongly agree, with higher scores indicating greater smoking urge). Example item: "I have a desire for a cigarette right now".
Electronic cigarette dependence | 12 months
  Levels of nicotine dependence associated with vaping will be assessed with the Penn State Electronic Cigarette Dependence Index (which consists a total of 9 questions, some multiple-choice questions, and some Yes/No questions; Higher scores indicate greater e-cigarette dependence).
Message effectiveness perceptions | 12 months
  The perceived message effectiveness of the anti-vaping PSAs will be evaluated using the Perceived Message Effectiveness scale, which is consisted of four items (1 = strongly disagree, 5 = strongly agree). Example items included "This message was convincing" and "Reading this message helped me feel confident about how to best deal with vaping."
Vaping intention | 12 months
  Vaping intention will be assessed through three self-reported items (1=very unlikely, 5=very likely). Example item: "I plan to vape or use e-cigarettes, even one or two puffs, in the next 6 months".
Smoking intention | 12 months
  Smoking intention will be assessed through three self-reported items (1=very unlikely, 5=very likely). Example item: "I plan to smoke cigarettes, even one or two puffs, in the next 6 months".
Self-report monthly other substance use severity | 12 months
  The frequency of other substance use will be assessed by the timeline follow-back measures. Specifically, participants will be asked to retrospectively estimate their daily use of other substances (including alcohol, marijuana, and other licit or illicit drug use) for the 7 days prior to the weekly survey date. The four weekly estimates will be averaged to create the monthly other substance use severity measure. The greater the number, the higher the other substance use severity in that month.

CONTACTS AND LOCATIONS:
Locations (1):
- UGA Bio-imaging Research Center, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
The proposed research is under the 500k threshold for required resource sharing. The PI and research team are committed to resource sharing; however, in the context of the proposed study, no plans are in place to make data available outside of the research team.